CLINICAL TRIAL: NCT03350503
Title: AcrySof IQ Toric A-Code Post-Market Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILV814-P001
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Cataract; Astigmatism
Keywords: phacoemulsification; intraocular lens; vision; toric
MeSH Terms: conditions — Cataract; Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Acrysof IQ Toric A-code IOL (Experimental): IOL implanted during cataract surgery
  Interventions: Device: AcrySof IQ Toric A-code IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: AcrySof IQ Toric A-code IOL — Intended to provide visual acuity, including astigmatism correction, over the lifetime of the cataract patient
  Other Names: Models SN6AT3, SN6AT4, SN6AT5
Procedure: Cataract surgery — Removal of cataractous lens and implantation of IOL

SUMMARY:
The purpose of this study is to clinically confirm the rotational stability of a modified AcrySof IQ toric intraocular lens (IOL) in a Japanese population.

DETAILED DESCRIPTION:
Patients will be examined pre-operatively to up to 3 years post-operatively. One eligible eye will be selected as a target eye for efficacy analysis. If both eyes are eligible, the eye in which the IOL is implanted first will be selected as the target eye.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cataracts with planned cataract removal by phacoemulsification
* Calculated lens power within the available range
* Able to sign informed consent and complete all study visits
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye conditions as specified in the protocol
* Uncontrolled glaucoma
* Pregnancy, current or planned
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Expert Clinical Project Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (4):
- Japan (4):
  - Alcon Investigative Site, Hiroshima, Hiroshima
  - Alcon Investigative Site, Hakodate, Hokkaido
  - Alcon Investigative Site, Miyakonojō, Miyazaki
  - Alcon Investigative Site, Saga, Saga-ken

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 4 investigative sites located in Japan.
Pre-assignment Details: Of the 125 subjects enrolled, 4 were exited as screen failures prior to implantation with the test article. This reporting group includes all subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye) (Safety Analysis Set).
Units Other Than Participants: eye
Groups:
- AcrySof IQ Toric A-code IOL: AcrySof IQ Toric A-code (SN6AT3 - SN6AT5) implanted in the study eye
Period: Overall Study
Arm/Group | AcrySof IQ Toric A-code IOL
Started | 121; 121 eye
Successful Implantation | 120; 120 eye
Implanted With SN6AT3 | 61; 61 eye
Implanted With SN6AT4 | 27; 27 eye
Implanted With SN6AT5 | 33; 33 eye
Completed | 104; 104 eye
Not Completed | 17; 17 eye
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 5
Not completed — Continuation impossible due to move | 4
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | Acrysof IQ Toric A-code IOL
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (7.0)
Age, Customized [Count of Participants; unit: Participants]
  Less than 60 years | 2
  60 to 69 years | 14
  70 to 79 years | 69
  Equal to or greater than 80 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 54
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 121
Region of Enrollment [Number; unit: participants]
  Japan | 121

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Absolute Value of Intraocular (IOL) Rotation (Visit 00 to Visit 4)
Description: IOL rotation was defined as the IOL axis difference between study visits. A photograph of the eye was taken, and IOL rotation was calculated as the angle between the toric mark on the IOL at Visit 4 and the reference point from Visit 00 (minimum 0 degrees, maximum 180 degrees). A lower value indicates greater IOL stability. No confirmatory hypothesis testing was conducted.
Time Frame: Visit 00 (Day 0 operative), Visit 4 (Day 120-180 postoperative)
Population: All Implanted Analysis Set: All eyes with successful test article implantation and measurable data at Visit 4.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eye
Arm/Group | Acrysof IQ Toric A-code IOL
Number analyzed (Participants) | 114
Number analyzed (eye) | 114
percentage of eyes
  Less than 10 degrees rotation | 99.1
  Greater than or equal to 10 degrees rotation | 0.9
  Less than 20 degrees rotation | 100.0
  Greater than or equal to 20 degrees rotation | 0.0
  Less than 30 degrees rotation | 100.0
  Greater than or equal to 30 degrees rotation | 0.0

2. Other Pre Specified Outcome: Percentage of Eyes With Absolute Value of IOL Rotation From Visit 00
Description: IOL rotation was defined as the IOL axis difference between study visits. A photograph of the eye was taken, and IOL rotation was calculated as the angle between the toric mark on the IOL at the specified visit and the reference point from Visit 00 (minimum 0 degrees, maximum 180 degrees). A lower value indicates greater IOL stability.
Time Frame: Visit 00 (Day 0 operative), Visit 00-A (Day 0, 1 +/- 0.5 hours postoperative), Visit 1 (Day 1-2 postoperative), Visit 2 (Day 7-14), Visit 3 (Day 30-60), Visit 4 (Day 120-180), Visit 5 (Day 330-420), Visit 6 (Day 630-780), Visit 7 (Day 990-1140)
Population: All Implanted Analysis Set: All eyes with successful test article implantation and measurable data at both visits.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eye
Groups:
- Visit 00 (Day 0 Operative); Visit 1 (Day 1-2 Postoperative); Visit 2 (Day 7-14 Postoperative); Visit 3 (Day 30-60 Postoperative); Visit 4 (Day 120-180 Postoperative); Visit 5 (Day 330-420 Postoperative); Visit 6 (Day 630-780 Postoperative); Visit 7 (Day 990-1140 Postoperative): AcrySof IQ Toric A-code (SN6AT3 - SN6AT5) implanted in the study eye
Arm/Group | Visit 00 (Day 0 Operative) | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 116 | 118 | 118 | 116 | 114 | 109 | 95 | 90
Number analyzed (eye) | 116 | 118 | 118 | 116 | 114 | 109 | 95 | 90
percentage of eyes
  Less than 10 degrees rotation | 100.0 | 100.0 | 99.2 | 99.1 | 99.1 | 99.1 | 98.9 | 100.0
  Greater than or equal to 10 degrees rotation | 0.0 | 0.0 | 0.8 | 0.9 | 0.9 | 0.9 | 1.1 | 0.0
  Less than 20 degrees rotation | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Greater than or equal to 20 degrees rotation | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Less than 30 degrees rotation | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Greater than or equal to 30 degrees rotation | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Other Pre Specified Outcome: Mean Absolute Value of IOL Rotation From Visit 00
Description: IOL rotation was defined as the IOL axis difference between study visits. A photograph of the eye was taken, and IOL rotation was calculated as the angle on the IOL at the specified visit and the reference point from Visit 00 (minimum 0 degrees, maximum 180 degrees). A lower value indicates greater IOL stability.
Time Frame: as for outcome 2
Population: All Implanted Analysis Set: All eyes with successful test article implantation and measurable data at both visits.
Measure: Mean (Standard Deviation); unit: degree
Units Other Than Participants: eye
Arm/Group | Visit 00 (Day 0 Operative) | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 116 | 118 | 118 | 116 | 114 | 109 | 95 | 90
Number analyzed (eye) | 116 | 118 | 118 | 116 | 114 | 109 | 95 | 90
degree | 2.11 (1.80) | 2.37 (1.96) | 2.22 (2.08) | 2.32 (2.14) | 2.30 (2.23) | 2.10 (2.08) | 2.31 (1.99) | 2.10 (2.06)

4. Other Pre Specified Outcome: Mean Uncorrected Distance Visual Acuity (UCDVA) by Visit
Description: Visual acuity (VA) was tested under well-lit conditions with no refractive correction in place using a decimal visual acuity chart set at 5 meters. VA was measured in "logarithm of the minimum angle of resolution" (logMAR), with 0.0 logMAR corresponding to 20/20 Snellen visual acuity, or normal distance eyesight. A negative value denotes better than 20/20 visual acuity.
Time Frame: Visit 0 (Preoperative), Visit 1 (Day 1-2 postoperative), Visit 2 (Day 7-14), Visit 3 (Day 30-60), Visit 4 (Day 120-180), Visit 5 (Day 330-420), Visit 6 (Day 630-780), Visit 7 (Day 990-1140)
Population: All Implanted Analysis Set: All eyes with successful test article implantation
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eye
Groups:
- Visit 0 (Preoperative): Prior to AcrySof IQ Toric A-code (SN6AT3 - SN6AT5) implanted in the study eye
Arm/Group | Visit 0 (Preoperative) | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 120 | 119 | 118 | 118 | 116 | 115 | 109 | 104
Number analyzed (eye) | 120 | 119 | 118 | 118 | 116 | 115 | 109 | 104
logMAR | 0.551 (0.368) | 0.087 (0.170) | 0.058 (0.156) | 0.040 (0.127) | 0.054 (0.149) | 0.045 (0.163) | 0.070 (0.157) | 0.086 (0.182)

5. Other Pre Specified Outcome: Mean Best Corrected Distance Visual Acuity (BCDVA) by Visit
Description: Visual acuity (VA) was tested under well-lit conditions with refractive correction in place using a decimal visual acuity chart set at 5 meters. VA was measured in "logarithm of the minimum angle of resolution" (logMAR), with 0.0 logMAR corresponding to 20/20 Snellen visual acuity, or normal distance eyesight. A negative value denotes better than 20/20 visual acuity.
Time Frame: as for outcome 4
Population: All Implanted Analysis Set: All eyes with successful test article implantation
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eye
Arm/Group | Visit 0 (Preoperative) | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 120 | 119 | 118 | 118 | 116 | 115 | 109 | 104
Number analyzed (eye) | 120 | 119 | 118 | 118 | 116 | 115 | 109 | 104
logMAR | 0.190 (0.163) | -0.030 (0.113) | -0.063 (0.088) | -0.080 (0.063) | -0.075 (0.099) | -0.085 (0.077) | -0.073 (0.080) | -0.069 (0.101)

6. Other Pre Specified Outcome: Mean Sub-Surface Nano Glistening (SSNG) Densitometry (Peak) by Visit
Description: Sub-surface nano glistening (SSNG) densitometry was measured as the IOL anterior surface light scattering densitometry using Pentacam or Pentacam HR. SSNG was measured in units specific to the device, with a higher number indicating a higher presence of SSNG. Peak value is the highest value in the IOL anterior surface light scattering densitometry.
Time Frame: Visit 1 (Day 1-2 postoperative), Visit 2 (Day 7-14), Visit 3 (Day 30-60), Visit 4 (Day 120-180), Visit 5 (Day 330-420), Visit 6 (Day 630-780), Visit 7 (Day 990-1140)
Population: All Implanted Analysis Set: All eyes with successful test article implantation
Measure: Mean (Standard Deviation); unit: arbitrary units
Units Other Than Participants: eye
Arm/Group | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 117 | 117 | 117 | 115 | 114 | 107 | 103
Number analyzed (eye) | 117 | 117 | 117 | 115 | 114 | 107 | 103
arbitrary units | 4.50 (0.70) | 4.55 (0.57) | 4.50 (0.55) | 4.48 (0.64) | 4.64 (0.78) | 4.82 (0.63) | 5.11 (0.76)

7. Other Pre Specified Outcome: Mean SSNG Densitometry (Area Analysis) by Visit
Description: Sub-surface nano glistening (SSNG) densitometry was measured as the IOL anterior surface light scattering densitometry using Pentacam or Pentacam HR. SSNG was measured in units specific to the device, with a higher number indicating a higher presence of SSNG. Area analysis value is an average value of the IOL anterior surface light scattering densitometry in a certain area.
Time Frame: as for outcome 6
Population: All Implanted Analysis Set: All eyes with successful test article implantation
Measure: Mean (Standard Deviation); unit: arbitrary units
Units Other Than Participants: eye
Arm/Group | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 117 | 117 | 117 | 115 | 114 | 107 | 103
Number analyzed (eye) | 117 | 117 | 117 | 115 | 114 | 107 | 103
arbitrary units | 4.07 (0.50) | 4.12 (0.47) | 4.08 (0.46) | 4.05 (0.42) | 4.19 (0.38) | 4.30 (0.41) | 4.45 (0.48)

8. Other Pre Specified Outcome: Number of Device Deficiencies
Description: A device deficiency was defined as an inadequacy of the medical device with respect to its identity, quality, durability, reliability, safety, or performance.
Time Frame: as for outcome 2
Population: Safety Analysis Set
Measure: Number; unit: device deficiency
Units Other Than Participants: eye
Groups:
- Overall: AcrySof IQ Toric A-code (SN6AT3 - SN6AT5) implanted in the study eye
Arm/Group | Overall
Number analyzed (Participants) | 121
Number analyzed (eye) | 121
device deficiency
  Broken IOL optic | 0
  Broken IOL haptic | 0
  IOL luxation | 0
  IOL dislocation | 0
  Other: IOL rotation | 2

9. Other Pre Specified Outcome: Percentage of Eyes With Glistening by Visit
Description: A slit lamp examination was conducted to determine the presence/absence of glistening particles on the implanted IOL. Glistening was reported by on a 4-point scale, where Grade 0 = no glistening; Grade 1 = mild glistening (50/mm3); Grade 2 = moderate glistening (100/mm3); and Grade 3 = severe glistening (200/mm3).
Time Frame: as for outcome 6
Population: Safety Analysis Set: All eyes with attempted implantation with the test article (successful or aborted after contact with the eye). Note: One subject implanted with the test article discontinued the study prior to the Visit 1 assessment.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eye
Arm/Group | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative)
Number analyzed (Participants) | 120 | 119 | 119 | 117 | 116 | 101 | 104
Number analyzed (eye) | 120 | 119 | 119 | 117 | 116 | 101 | 104
percentage of eyes
  Grade 0 | 100.0 | 100.0 | 100.0 | 88.0 | 68.1 | 59.4 | 49.0
  Grade 1 | 0.0 | 0.0 | 0.0 | 9.4 | 20.7 | 21.8 | 27.9
  Grade 2 | 0.0 | 0.0 | 0.0 | 2.6 | 7.8 | 13.9 | 15.4
  Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 3.4 | 5.0 | 7.7

10. Other Pre Specified Outcome: Number of Eyes With Posterior Capsule Opacification (PCO) by Visit
Description: A slit lamp examination was performed to evaluate the eye for posterior capsule opacification (that is, the thickening, opacification and clouding of the posterior lens capsule). The presence or absence of PCO was recorded. Clinical significance was determined by the investigator.
Time Frame: Visit 1 (Day 1-2 postoperative), Visit 2 (Day 7-14), Visit 3 (Day 30-60), Visit 4 (Day 120-180), Visit 5 (Day 330-420), Visit 6 (Day 630-780), Visit 7 (Day 990-1140), Unscheduled Visits between Visit 1 and Visit 7
Population: as for outcome 9
Measure: Number; unit: eye
Units Other Than Participants: eye
Groups:
- Unscheduled Visits Between Visit 1 and Visit 7; Visit 1 Through Visit 7 Cumulative: AcrySof IQ Toric A-code (SN6AT3 - SN6AT5) implanted in the study eye
Arm/Group | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative) | Unscheduled Visits Between Visit 1 and Visit 7 | Visit 1 Through Visit 7 Cumulative
Number analyzed (Participants) | 120 | 119 | 119 | 117 | 116 | 105 | 104 | 21 | 120
Number analyzed (eye) | 120 | 119 | 119 | 117 | 116 | 105 | 104 | 21 | 120
eye
  None | 120 | 118 | 112 | 105 | 100 | 79 | 66 | 16 | 74
  Clinically nonsignificant | 0 | 1 | 7 | 12 | 16 | 26 | 34 | 0 | 39
  Clinically significant | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
  Clinically significant requiring Nd:YAG laser treatment | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 5

11. Other Pre Specified Outcome: Number of Eyes Receiving Nd:YAG Laser Treatment for Posterior Capsule Opacification (PCO) by Visit
Description: A slit lamp examination was performed to evaluate the eye for posterior capsule opacification (that is, the thickening, opacification and clouding of the posterior lens capsule). A neodymium-doped yttrium aluminum garnet (Nd:YAG) laser was used to treat posterior capsule opacification, with treatment determined by the investigator. The presence or absence of Nd:YAG laser treament was recorded.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Number; unit: eye
Units Other Than Participants: eye
Arm/Group | Visit 1 (Day 1-2 Postoperative) | Visit 2 (Day 7-14 Postoperative) | Visit 3 (Day 30-60 Postoperative) | Visit 4 (Day 120-180 Postoperative) | Visit 5 (Day 330-420 Postoperative) | Visit 6 (Day 630-780 Postoperative) | Visit 7 (Day 990-1140 Postoperative) | Unscheduled Visits Between Visit 1 and Visit 7 | Visit 1 Through Visit 7 Cumulative
Number analyzed (Participants) | 120 | 119 | 119 | 117 | 116 | 110 | 104 | 32 | 120
Number analyzed (eye) | 120 | 119 | 119 | 117 | 116 | 110 | 104 | 32 | 120
eye
  No | 120 | 119 | 119 | 117 | 116 | 110 | 103 | 29 | 116
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the duration of individual participation (up to 990-1140 days).
Description: Adverse Events were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. This analysis population includes all eyes with attempted implantation of the test article (successful or aborted after contact with the eye).
Groups:
- Acrysof IQ Toric A-code IOL: AcrySof IQ Toric A-code (SN6AT3 - SN6AT5) implanted unilaterally
Arm/Group | Acrysof IQ Toric A-code IOL
All-Cause Mortality (participants affected / at risk) | 4/121
Serious Adverse Events (participants affected / at risk) | 15/121
Other Adverse Events (participants affected / at risk) | 7/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acrysof IQ Toric A-code IOL (N=121)
Cerebral infarction (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Haemmorhoids (Gastrointestinal disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Dermatochalasis (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acrysof IQ Toric A-code IOL (N=121)
Posterior capsule opacification (Eye disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT03350503/Prot_002.pdf
  • Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03350503/SAP_003.pdf